CLINICAL TRIAL: NCT06979804
Title: A Comparison of Outcomes After Anterior Cruciate Ligament (ACL) or Anterior Cruciate Ligament and Meniscus (ACL+Meniscus) Surgery Using Semiconductor Fabric Products: A Randomized, Double-Blinded, Placebo-Controlled Prospective Clinical Study
Brief Title: A Comparison of Outcomes After Anterior Cruciate Ligament (ACL) or Anterior Cruciate Ligament and Meniscus (ACL+Meniscus) Surgery Using Semiconductor Fabric Products
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Illinois Center for Orthopaedic Research and Education (Other)
Collaborators: INCREDIWEAR HOLDINGS, INC. (Industry)
Responsible Party: Principal Investigator, Ronak M. Patel, Sports Medicine Orthopedic Surgeon, Illinois Center for Orthopaedic Research and Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12178
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: ACL Reconstruction; Meniscus Tears; Anterior Cruciate Ligament Rupture
Keywords: ACL; Meniscus tear; ACL tear; Compression sleeve; Semiconductor fabric; ACL reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Control Group (No Intervention): This arm of the study involves the control group who will receive the standard of care.
- Semiconducting Fabric Sleeve Group (Active Comparator): This group will be receiving semiconducting fabric sleeve to be worn post-operatively.
  Interventions: Device: Semiconducting fabric sleeves
- Placebo Group (Placebo Comparator): This group receives a look-alike sleeve that contains no semiconductor material.
  Interventions: Device: Non-semiconducting fabric sleeves

INTERVENTIONS:
Device: Semiconducting fabric sleeves — This intervention includes semiconductor embedded sleeves that patients will wear for 4 months post-operatively.
  Arms: Semiconducting Fabric Sleeve Group
Device: Non-semiconducting fabric sleeves — This intervention includes sleeves absent of semiconductors that will be worn for 4 months post-operatively.
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to determine the effect of semiconductor sleeves on the treatment of Anterior Cruciate Ligament (ACL) or Anterior Cruciate Ligament and Meniscus (ACL+Meniscus) arthroscopic surgery. The effect of the sleeves will be analyzed through patient reported and clinically measured outcomes. The main questions it aims to answer are:

* Do the semiconductor sleeves improve the functional outcomes compared to the placebo?
* Will patients experience improved functional outcomes in a shorter period of time compared to the placebo?

Researchers will compare semiconductor fabric sleeves to a placebo (a look-alike sleeve that contains no semiconductor material) to see if the semiconductor fabric better treats ACL and ACL+meniscus surgical patients.

Participants will:

* Wear semiconductor or placebo leg sleeve for 4 weeks and knee sleeve for the following 12 weeks
* Complete patient reported outcome surveys

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ACL or ACL+Meniscus surgery
* Age 16 - 65
* Patients with Body Mass Index (BMI) <40
* Patients who are willing and able to adhere to follow-up schedule and protocol guidelines.
* Patients who are willing and able to sign corresponding research subject consent/assent form.

Exclusion Criteria:

* Patient has a history of neurological conditions, including multiple sclerosis or Parkinson's disease
* Patient has severe medical condition, including recent myocardial infarction, unstable angina, heart failure, severe anemia
* Patient has had prior surgical treatment of the knee in the last 5 years or injection treatment(s) in the last 6 months
* Patient has chronic pain conditions unrelated to knee condition
* Patient has auto-immune or auto-inflammatory diseases
* Patient has poorly controlled diabetes (HgA1c > 7.5)
* Patient has BMI > 39.9
* Patient has varicosities on the operative leg
* Patient has severe peripheral artery disease (ABI < 0.6)
* Patient is considered a pain management patient
* Patient has had previous blood clots or stroke
* Patient has used tobacco within the last 90 days
* Patient is not within the ages of 16-65
* Patient has an active infection (local or systemic), or an open (non-surgical) wound in the areas of product application
* Patient is unwilling or unable to sign the corresponding research subject consent/assent form
* Patient meets any other criteria or has any other condition that, in the opinion of the investigator, would prevent them from completing the study or that, in the opinion of the investigator, would confound study results.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Range of motion | 1 year
  Measured extension and flexion values using a goniometer at baseline, 2 weeks, 6 weeks, 3 months, 6 months, and 1 year time points

SECONDARY OUTCOMES:
Effusion Measurements | 1 year
  Effusion is measured by taking the circumference using a soft measuring tape at the following points:
  1. Mid thigh: distance from palpation of Anterior Superior Iliac Spine (ASIS) to superior pole of patella, divided in half. (cm)
  2. Knee: midpoint of the patella. (cm)
  3. Mid calf: distance from top of fibular head to bottom of lateral malleolus, divided in half. (cm)
Secondary Outcome Measures using Validated patient-reported outcome tools questionnaires | 1 year
  Visual Analog Scale (VAS) - assess pain, It is a 0-100 scale. A higher score indicates greater pain intensity.
Secondary Outcome Measures using Validated patient-reported outcome tools questionnaires | 1 year
  International Knee Documentation Committee (IKDC) - assesses symptoms and function in daily living activities
Secondary Outcome Measures using Validated patient-reported outcome tools questionnaires | 1 year
  Knee Single Assessment Numeric Evaluation (SANE) - assess knee function on a scale of 0 to 100, with 100 representing normal function
Secondary Outcome Measures using Validated patient-reported outcome tools questionnaires | 1 year
  Tegner Activity Scale - assesses work/sport activities level on a scale of 0 to 10, with 0 representing sick leave and 10 representing elite competitive sports.
Secondary Outcome Measures using Validated patient-reported outcome tools questionnaires | 1 year
  Lysholm Scale - assesses pain, instability, locking, swelling, limp, stair-climbing, squatting, and use of support after ligament surgery on a scale of 0 to 100.
Secondary Outcome Measures using Validated patient-reported outcome tools questionnaires | 1 year
  Knee injury and Osteoarthritis Outcome Score Jr (KOOS Jr) - assess five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. It is a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems

CONTACTS AND LOCATIONS:
Locations (1):
- Illinois Bone and Joint Institute, Westmont, Illinois, United States

REFERENCES:
- [Background] O'Riordan SF, Bishop DJ, Halson SL, Broatch JR. Do Sports Compression Garments Alter Measures of Peripheral Blood Flow? A Systematic Review with Meta-Analysis. Sports Med. 2023 Feb;53(2):481-501. doi: 10.1007/s40279-022-01774-0. Epub 2023 Jan 9. PMID 36622554
- [Background] Leung TK. In Vitro and In Vivo Studies of the Biological Effects of Bioceramic (a Material of Emitting High Performance Far-Infrared Ray) Irradiation. Chin J Physiol. 2015 Jun 30;58(3):147-55. doi: 10.4077/CJP.2015.BAD294. PMID 26014120
- [Background] Justice TE, Jacob PB. Non-compressive sleeves versus compression stockings after total knee arthroplasty: A prospective pilot study. J Orthop. 2023 Nov 24;49:102-106. doi: 10.1016/j.jor.2023.11.044. eCollection 2024 Mar. PMID 38094981